CLINICAL TRIAL: NCT05898438
Title: The Role of Gut Microbiota in Children With Epilepsy Following Ketogenic Diet
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Collaborators: Harokopio University (Other)
Responsible Party: Principal Investigator, Sofia D. Zouganeli, Principal Investigator, Attikon Hospital
Other Study IDs: ΕΒΔ620/30-09-2019
Record Dates: First submitted 2023-04-10; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Epilepsy
Keywords: ketogenic diet; epilepsy; children; gut microbiota
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The role of human microbiota in neurological disorders via the "microbiota-gut-brain axis" is recently gaining increased attention due to the knowledge that gut microorganisms are involved in multiple gut and brain functions and metabolic pathways. The hypothesis of the present investigation is that changes of gut microbiota and their metabolic products may be a mechanism of the effectiveness of ketogenic diet in epilepsy.

The aim of the present study is to investigate the changes of gut microbiota induced by the ketogenic diet and if certain populations of microorganisms are associated with better seizure control in epileptic children.

This is a non-interventional study that will include epileptic children 2-18 years old eligible for ketogenic diet. The gut microbiome of participants will be examined in stools before and three months after the implementation of an olive oil- based ketogenic diet therapy. One of the participants' parents will also be included providing fecal sample for the examination of gut microbiome.

DETAILED DESCRIPTION:
The high-fat, adequate protein, low-carbohydrate ketogenic diet (KD) has successfully been used in the treatment of drug resistant epilepsy (DRE) in children since 1920's. The classical KD, with fat to carbohydrate plus protein ratio of 3 or 4:1, as well as less restrictive forms such as Modified Atkins Diet (MAD) or Low Glycemic Index Therapy (LGIT), have been proved to be effective in reducing seizures more than 50% in many patients with low response to more than two antiepileptic drugs (AEDs). Apart from a great number of epileptic syndromes, metabolic conditions like GLUT I-Glucose Transporter I - Deficiency Syndrome and Pyruvate Dehydrogenase Deficiency Syndrome seem to be especially responsive to KD.

The role of human microbiota in neurological disorders via the "microbiota-gut-brain axis" with gut microorganisms getting involved in multiple gut and brain functions and metabolic pathways has recently gained attention .The changes of gut microbiota by the low carbohydrate and low fibre ketogenic diet seem to have an impact on its effectiveness in epilepsy control. Furthermore, metabolic products of gut microorganisms such as SCFAs, apart from producing energy, are implicated in inflammatory pathways and are directly affected by the low fibre - carbohydrate content of the ketogenic diet.

The small number of studies so far confirm the role of gut microbiome in seizure control without specifying the exact mechanisms yet. The aim of the present study is to further investigate how gut microbiota and the metabolic products of microorganisms are implicated in the effectiveness of ketogenic diet therapy in epileptic children.

The study will include epileptic children 2-18 years old eligible for ketogenic diet according to ILAE. The gut microbiome of participants will be examined at the beginning of the study and three months after following an olive-oil based ketogenic diet therapy. One of the participants' parents will also be included, providing fecal samples for the examination of gut microbiome. A written informed consent will be provided by all the participants or care givers.

This is a prospective, non-interventional study which will be held in the Department of Pediatric Neurology, 3d Pediatric Clinic, Attikon Athens University Hospital, in collaboration with the Department of Nutrition and Dietetics, Harokopio University. The study has received approval by the Ethics Committee and the Scientific Board of the Attikon Athens University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* type of epilepsy requiring ketogenic diet (drug-resistant epilepsy or Glut 1 DS or PDHD)
* eligibility for ketogenic diet according to ILAE
* no antibiotic intake for at least 2 months before the beginning of the study
* no probiotics or prebiotics intake for at least 2 weeks before the beginning of the study

Exclusion Criteria:

- systematic diseases (e.g. inflammatory bowel disease, cancer, autoimmune and cardiometabolic diseases)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with epilepsy visiting Pediatric Neurology Department of 3rd Pediatric Clinic, Attikon Athens University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of epileptic seizures frequency | 3 months
  Recording of number of seizures per week/month Recording the ratio of epileptic seizures change e.g. decrease >50%, decrease 50-90%, decrease >90%
Changes in electroengephalographic activity | 3 months
  Subjective assessment of neurophysiologist depending on the diagnosis of each patient's epileptic syndrome.
  Measurement of Spike Wave Index (%) in Electrical Status Epilepticus During Slow-wave Sleep (ESES)

SECONDARY OUTCOMES:
Alterations in gut microbiota | 3 months
  alterations in specific gut microbial populations (quantitative real time PCR)
Changes in gut microbial metabolites | 3 months
  Short Chain Fatty Acids quantification (gas chromatography)

CONTACTS AND LOCATIONS:
Overall Officials: Argirios Dinopoulos, Professor, Study Chair — 3rd Pediatric Clinic, Attikon Athens University Hospital
Locations (1):
- Attikon Athens University Hospital, Athens, Haidari, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olson CA, Vuong HE, Yano JM, Liang QY, Nusbaum DJ, Hsiao EY. The Gut Microbiota Mediates the Anti-Seizure Effects of the Ketogenic Diet. Cell. 2018 Jun 14;173(7):1728-1741.e13. doi: 10.1016/j.cell.2018.04.027. Epub 2018 May 24. PMID 29804833
- [Background] Xie G, Zhou Q, Qiu CZ, Dai WK, Wang HP, Li YH, Liao JX, Lu XG, Lin SF, Ye JH, Ma ZY, Wang WJ. Ketogenic diet poses a significant effect on imbalanced gut microbiota in infants with refractory epilepsy. World J Gastroenterol. 2017 Sep 7;23(33):6164-6171. doi: 10.3748/wjg.v23.i33.6164. PMID 28970732
- [Background] Zhang Y, Zhou S, Zhou Y, Yu L, Zhang L, Wang Y. Altered gut microbiome composition in children with refractory epilepsy after ketogenic diet. Epilepsy Res. 2018 Sep;145:163-168. doi: 10.1016/j.eplepsyres.2018.06.015. Epub 2018 Jun 28. PMID 30007242
- [Background] Lindefeldt M, Eng A, Darban H, Bjerkner A, Zetterstrom CK, Allander T, Andersson B, Borenstein E, Dahlin M, Prast-Nielsen S. The ketogenic diet influences taxonomic and functional composition of the gut microbiota in children with severe epilepsy. NPJ Biofilms Microbiomes. 2019 Jan 23;5(1):5. doi: 10.1038/s41522-018-0073-2. eCollection 2019. PMID 30701077
- [Background] Tagliabue A, Ferraris C, Uggeri F, Trentani C, Bertoli S, de Giorgis V, Veggiotti P, Elli M. Short-term impact of a classical ketogenic diet on gut microbiota in GLUT1 Deficiency Syndrome: A 3-month prospective observational study. Clin Nutr ESPEN. 2017 Feb;17:33-37. doi: 10.1016/j.clnesp.2016.11.003. Epub 2016 Dec 18. PMID 28361745
- [Background] Gong X, Cai Q, Liu X, An D, Zhou D, Luo R, Peng R, Hong Z. Gut flora and metabolism are altered in epilepsy and partially restored after ketogenic diets. Microb Pathog. 2021 Jun;155:104899. doi: 10.1016/j.micpath.2021.104899. Epub 2021 Apr 21. PMID 33894293
- [Background] Peng A, Qiu X, Lai W, Li W, Zhang L, Zhu X, He S, Duan J, Chen L. Altered composition of the gut microbiome in patients with drug-resistant epilepsy. Epilepsy Res. 2018 Nov;147:102-107. doi: 10.1016/j.eplepsyres.2018.09.013. Epub 2018 Sep 24. PMID 30291996